CLINICAL TRIAL: NCT02103803
Title: Assessing Eye Tracking Features Following Sports-Related Concussion
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Lee Family Foundation (Unknown)
Responsible Party: Principal Investigator, Jamie M. Bogle, Au.D., Ph.D., Senior Associate Consultant, Mayo Clinic
Other Study IDs: 13-009632
Record Dates: First submitted 2014-03-19; First posted 2014-04-04 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Traumatic Brain Injury
Keywords: concussion; sports-related concussion; mild traumatic brain injury (mTBI); eye tracking; oculometrics
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This proposal aims to describe the oculometric features present during King-Devick (K-D) testing for subjects who experienced sports-related concussion. The investigators aim to better describe the underlying oculomotor anomalies present in this cohort that lead to increased K-D test time. Understanding these anomalies will allow for better understanding of the effects of sports-related concussion and may provide a rapid and reliable metric for diagnosing concussion as well as monitoring long-term recovery.

DETAILED DESCRIPTION:
This proposal aims to describe the oculometric features present during K-D testing for subjects who experienced sports-related concussion. The investigators aim to better describe the underlying oculomotor anomalies present in this cohort that lead to increased K-D test time. Understanding these anomalies will allow for better understanding of the effects of sports-related concussion and may provide a rapid and reliable metric for diagnosing concussion as well as monitoring long-term recovery.

The main objectives include:

1. Describing the oculometric deficits present in subjects with acute sports-related concussion.
2. Analyzing and quantifying the oculometric changes that occur during subject recovery.
3. Identifying possible oculometric features as potential biomarkers that may lead to reliable, rapid method for recognizing acute concussion.

ELIGIBILITY:
Inclusion criteria:

* Over the age of 8 years, and able to provide informed consent / assent.
* Have documented diagnosis of sports-related concussion within two weeks of the event.
* Currently demonstrating post-concussion symptoms.

Exclusion criteria:

- Alcohol consumption within 48 hours of evaluation.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Twenty subjects with diagnosed concussion will be recruited from the adolescent and adult population seen in the Comprehensive Concussion Program at Mayo Clinic Arizona.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2014-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in time to complete King-Devick Test | Baseline to 4 weeks
  The King-Devick Test (K-D Test) is a two-minute test that requires an athlete to read single digit numbers displayed. Subjects will be seated in front of a computer screen and eye tracking device connected to the computer. The eye tracking device consists of infrared cameras, which captured eye movements by tracking the reflections of infrared reference lights on the subjects' retinas. Before the start of the experiment, they will begin by watching a moving target on the computer screen to calibrate the system. Then, the subject completes a computerized version of the K-D test. The K-D test requires that the subject rapidly read aloud the numbers presented on the three test cards. Reading the three test cards requires less than two minutes to complete. The number of errors will be counted. Oculometric data will be collected during the test and analyzed offline. The total time required to complete all three test cards is the completion time for the entire K-D test.

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Pradhan, PhD, Principal Investigator — Mayo Clinic; Jan Stepanek, MD, Principal Investigator — Mayo Clinic; Jamie Bogle, AuD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States